CLINICAL TRIAL: NCT02035722
Title: A Visual Approach to Reducing Anxiety and Improving Knowledge Transfer for Patients Receiving Intravitreal Injections
Brief Title: Intravitreal Injections-related Anxiety
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHN-110463AE
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (No Intervention): AMD-related information is not given to patients randomized to the control group.
- Video materials (Active Comparator): Educational materials are presented in through a video (audio and visual)
  Interventions: Behavioral: Video
- Print materials (Active Comparator): Educational materials are presented in the format of printed brochure (visual)
  Interventions: Behavioral: Printed materials

INTERVENTIONS:
Behavioral: Printed materials — AMD-related information is presented to patients in the form of a brochure (i.e. printed materials)
  Arms: Print materials
Behavioral: Video — AMD-related information is presented as in the form of a video
  Arms: Video materials

SUMMARY:
Intravitreal injection of Ranibizumab (Lucentis, Genentech) is clinically indicated for patients with wet age-related macular degeneration (AMD) An disadvantage of this technique is the anxiety and discomfort which patients often experience due to the idea of "getting a needle in the eye". In addition, a recent case study indicated the importance of patient education in achieving positive outcomes from intravitreal injections of anti-vascular endothelial growth factor (VEGF) agents. The purpose of our study is to determine whether visual education on AMD and intravitreal injection can reduce patients' anxiety prior to the treatment, and lessen the impact of socioeconomical status on their understanding of the treatment and prognosis.

DETAILED DESCRIPTION:
The use of intravitreal injections of Ranibizumab (Lucentis, Genentech) is becoming increasing common for the management of age-related macular degeneration (AMD). It is therefore important to acknowledge and address patients' anxiety due to anticipated discomfort from the idea of "getting a needle in the eye". In addition, visual provision of information at diagnosis concerning long-term treatment expectation may enhance the informed consent process. The use of visual aids may also accommodate patients of different educational background when presented with new and complex treatment information. The purpose of our study is to determine whether visual education on AMD and intravitreal injection can reduce patients' anxiety prior to the treatment, and lessen the impact of socioeconomical status on their understanding of the treatment and prognosis. Although this tool will be developed in the context of injection-requiring retinal diseases, it has applications in the care of disease requiring long-term treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* AMD patients requiring intravitreal injections

Exclusion Criteria:

* Unable to read or comprehend English
* Any contraindications to intravitreal injections, such as IOP elevations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Anxiety | Cross-sectional study, where questionnaires will be completed on the same day of clinic visit.

SECONDARY OUTCOMES:
Knowledge of AMD | Cross-sectional study, where questionnaires will be completed on the same day of clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Wai-Ching Lam, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada